CLINICAL TRIAL: NCT06960031
Title: Added Value of PET/CT in Assessment of Hepatocellular Malignancy Post Radiofrequency Ablation
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Naglaa Samy Fahmy Abou Taira, Lecturer of Diagnostic Radiology and Medical Imaging, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR1162/3/25
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: PET/CT; Hepatocellular Malignancy; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PET/CT: Hybrid positron emission tomography (PET) and computed tomography (CT) images will be performed using Philips hybrid system equipped with a 16 MDCT scanner.
  The whole-body PET images from the skull vault down to the knee will be performed using several bed positions acquisition, each bed is approximately 15cm axial filed with 4mm special resolution. The time of acquisition of the emission scan is about 2 min for each bed, with a total time range between 12 and 17 min.
  Interventions: Other: PET/CT technique

INTERVENTIONS:
Other: PET/CT technique — Hybrid positron emission tomography (PET) and computed tomography (CT) images will be performed using Philips hybrid system equipped with a 16 MDCT scanner.
  The whole-body PET images from the skull vault down to the knee will be performed using several bed positions acquisition, each bed is approximately 15cm axial filed with 4mm special resolution. The time of acquisition of the emission scan is about 2 min for each bed, with a total time range between 12 and 17 min.

SUMMARY:
This study aims to assess the residual tumoral activity versus the well ablation of اepatocellular carcinoma (HCC) post radiofrequency ablation.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary liver malignancy and is a leading cause of cancer-related death worldwide. It is the third most common cause of death of cancer worldwide, also the sixth and fourth common cancer in worldwide and Egypt, respectively.

Radiofrequency ablation (RFA) is a technique that is recently developed for the ablation of liver tumours. It converts radio frequency waves into thermal energy, causing coagulation necrosis of the tumours. It has attracted great interest in recent years because of the excellent response rate with little morbidity. Compared with other local ablative modalities, RFA has been shown to be safer and more effective.

Positron emission tomography (PET) with 18F-fluoro-2- deoxy-D-glucose (18F-FDG) is a functional imaging tool that provides metabolic information of the lesion. It is effective for diagnosis, monitoring therapy and detection of recurrent tumours of various cancers because of its high sensitivity and specificity. However, it is less successful in the detection of primary HCC because of variable uptake. Even though the value of 18F-FDG PET for the detection of primary HCC remains controversial, 18F-FDG PET would seem to be appropriate for the follow-up of liver tumours.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 75 years.
* Both sexes.
* Patients with hepatocellular carcinoma (HCC) and underwent radiofrequency ablation (RFA) .

Exclusion Criteria:

* Patients with past history of contrast allergy.
* Patients with blood glucose level >200 mg/dl at the time of the study.
* High serum creatinine> 2 mg / dl.
* Small lesions < 10 mm.
* Well differentiated hepatocellular carcinoma (HCC) lesions by pathology.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study will be carried out on 70 patients with hepatocellular malignancy at Tanta University Hospitals for a period from April 2025 to September 2025 after approval from institutional ethical committee.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of fluoro-2- deoxy-D-glucose (FDG) Positron emission tomography (PET) /computed tomography (CT) to predict hepatocellular carcinoma (HCC) | From 1 month to 3 months post radiofrequency ablation
  Sensitivity of fluoro-2- deoxy-D-glucose (FDG) Positron emission tomography (PET) /computed tomography (CT) to predict hepatocellular carcinoma (HCC) will be measured.

SECONDARY OUTCOMES:
The value of fluoro-2- deoxy-D-glucose (FDG) Positron emission tomography (PET) /computed tomography (CT) | From 1 month to 3 months post radiofrequency ablation
  The value of fluoro-2- deoxy-D-glucose (FDG) Positron emission tomography (PET) /computed tomography (CT)T in post radiofrequency ablation (RFA) follow up (Specificity, PPV, NPV, Accuracy) will be recorded.
Serum Alpha-Fetoprotein (AFP) level | From 1 month to 3 months post radiofrequency ablation
  Serum Alpha-Fetoprotein (AFP) level will be recorded
Mean diameter of ablated area and the mean of Liver standardized uptake value (SUvmax) . | From 1 month to 3 months post radiofrequency ablation
  Semi-quantitative evaluation: is including the SUvmax (standardized uptake value) and the ratio of tumour SUvmax to normal liver SUv mean (TSUvmax/LSUvmean) will be evaluated by drawing region of interest (ROI) encircling the tumour and drawing ROI for normal liver uptake.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author